CLINICAL TRIAL: NCT03380429
Title: An Open Label, Randomised, Parallel Group Clinical Study to Evaluate the Effect of the Connected Inhaler System (CIS) on Adherence to Relvar/Breo ELLIPTA Therapy, in Asthmatic Subjects With Poor Control
Brief Title: A Clinical Study to Evaluate the Effect of the Connected Inhaler System (CIS) on Adherence to Maintenance Therapy in Poorly Controlled Asthmatic Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 207040; 2017-002266-45 (EudraCT Number)
Record Dates: First submitted 2017-12-15; First posted 2017-12-21 (Actual); Results first posted 2020-02-05 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-03

CONDITIONS: Asthma
Keywords: Connected Inhaler System; Metered Dose Inhaler; ELLIPTA; RELVAR/BREO; Dry Powder Inhaler; Salbutamol; Asthma
MeSH Terms: conditions — Asthma | interventions — Albuterol

STUDY DESIGN:
Intervention Model Description: Eligible subjects will receive RELVAR/BREO maintenance therapy via ELLIPTA DPI and salbutamol rescue medication via MDI. Clip-on sensors will be attached to both inhalers which will provide data on maintenance therapy and rescue medication use to the subjects and their HCP. Subjects will be randomized into five treatment arms in a ratio of 1:1:1:1:1 depending on whether the data, from RELVAR/BREO ELLIPTA or RELVAR/BREO ELLIPTA and salbutamol MDI, is fed back to the subject or subject and HCP, or not at all.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (5):
- Data on Maintenance use supplied to Subject and HCP (Experimental): Eligible subjects will receive RELVAR/BREO maintenance therapy via ELLIPTA DPI and salbutamol rescue medication via MDI with sensors attached to both inhalers. Information from sensor attached to RELVAR/BREO ELLIPTA will be fed back to the subject via an app on smart phone and to the subject's HCP via an online dashboard.
  Interventions: Drug: RELVAR/BREO; Drug: Salbutamol; Device: Smart phone app; Device: HCP Dashboard; Device: Sensors
- Data on Maintenance use supplied to Subject (Experimental): Eligible subjects will receive RELVAR/BREO maintenance therapy via ELLIPTA DPI and salbutamol rescue medication via MDI with sensors attached to both inhalers. Information from sensor attached to RELVAR/BREO ELLIPTA will be fed back to the subject via an app on smart phone.
  Interventions: Drug: RELVAR/BREO; Drug: Salbutamol; Device: Smart phone app; Device: Sensors
- Data on Maintenance and Rescue use supplied to Subject and HCP (Experimental): Eligible subjects will receive RELVAR/BREO maintenance therapy via ELLIPTA DPI and salbutamol rescue medication via MDI with sensors attached to both inhalers. Information from sensors attached to RELVAR/BREO ELLIPTA and salbutamol MDI will be fed back to both subject and HCP. The data will be fed back to the subject through an app and to HCP through an online dashboard.
  Interventions: Drug: RELVAR/BREO; Drug: Salbutamol; Device: Smart phone app; Device: HCP Dashboard; Device: Sensors
- Data on Maintenance and Rescue use supplied to Subject (Experimental): Eligible subjects will receive RELVAR/BREO maintenance therapy via ELLIPTA DPI and salbutamol rescue medication via MDI with sensors attached to both inhalers. Information from sensors attached to RELVAR/BREO ELLIPTA and salbutamol MDI will be fed back to subject through an app.
  Interventions: Drug: RELVAR/BREO; Drug: Salbutamol; Device: Smart phone app; Device: Sensors
- No data supplied to Subject or HCP (Active Comparator): Eligible subjects will receive RELVAR/BREO maintenance therapy via ELLIPTA DPI and salbutamol rescue medication via MDI with sensors attached to both inhalers. Subjects will be provided with a home hub through which their data will be uploaded during the study but the subjects and their HCP will not be able to view the data.
  Interventions: Drug: RELVAR/BREO; Drug: Salbutamol; Device: Sensors

INTERVENTIONS:
Drug: RELVAR/BREO — RELVAR/BREO will be available at doses of 100/25 micrograms (µg) and 200/25 µg to be administered via ELLIPTA DPI. Subjects will be administered one inhalation of RELVAR/BREO once daily.
Drug: Salbutamol — Salbutamol will be available at a dose of 100 µg to be administered via MDI. Subjects will be administered salbutamol as and when required.
Device: Smart phone app — Subjects will be required to download an app associated with sensor on their smartphone. The sensors attached to the inhalers will be connected to the smartphone via Bluetooth.
  Arms: Data on Maintenance and Rescue use supplied to Subject; Data on Maintenance and Rescue use supplied to Subject and HCP; Data on Maintenance use supplied to Subject; Data on Maintenance use supplied to Subject and HCP
Device: HCP Dashboard — The information from sensors will be reviewed by the HCP via an online dashboard.
  Arms: Data on Maintenance and Rescue use supplied to Subject and HCP; Data on Maintenance use supplied to Subject and HCP
Device: Sensors — Clip-on sensors will be fitted to electronically record the actuation data.

SUMMARY:
GlaxoSmithKline (GSK) in collaboration with Propeller Health has developed a sensor, which can clip on to the ELLIPTA® dry powder inhaler (DPI) and monitor the time and date that the ELLIPTA DPI cover is fully opened and closed. Additionally, a sensor will be attached to the rescue medication metered dose inhaler (MDI). The data from both sensors will be fed back to the subject via an application (app) on smart phone and will be reviewed by the subject's health care professional (HCP) via an online dashboard. The sensors, app, dashboard and systems to provide data comprise the CIS. This study will be the first to evaluate the effect of CIS on adherence to maintenance therapy in subjects with uncontrolled asthma. This is an open-label, randomized, parallel group study in asthmatic subjects currently on a fixed dose inhaled corticosteroid (ICS)/long-acting beta 2 agonist (LABA) maintenance therapy. Eligible subjects will receive RELVAR®/BREO® maintenance therapy via ELLIPTA DPI and salbutamol rescue medication via MDI with sensors attached to both inhalers during the run-in period, which may last for up to 3 months. Eligible subjects will then be randomized into five treatment arms depending on whether the data, from RELVAR/BREO ELLIPTA or RELVAR/BREO ELLIPTA and salbutamol MDI, is fed back to the subject or subject and HCP, or not at all. The treatment period for the study is approximately 6 months and there will be a follow-up period one week post last visit. The total duration of a subject in the study will be approximately 9 months. RELVAR, BREO and ELLIPTA are registered trademarks of GlaxoSmithKline group of companies.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 years or older, at the time of signing the informed consent.
* Subjects with documented physician diagnosis of asthma as their primary respiratory disease.
* ACT score <20 at screening visit.
* Non-smokers (never smoked or not smoking for >6 months with <10 pack years history (Pack years = [cigarettes per day smoked/20] multiplied by number of years smoked).
* Male or female subjects will be included. A female subject is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies: (i) Not a woman of childbearing potential (WOCBP). (ii) A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 5 days] after the last dose of study treatment.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and protocol.
* Subject understands and is willing, able, and likely to comply with study procedures and restrictions.
* Subject must be able to read in a language supported by the smart phone app in their region.
* Subject must have been on maintenance therapy (Fixed dose combination ICS/LABA) for 3 months, cannot have changed dose in the month prior to screening and be able to change to an equivalent dose of RELVAR/BREO for the duration of the study. Other background asthma medication such as anti-leukotrienes and oral corticosteroids are permitted provided the dose has been stable for 1 month prior to screening.
* Subject must be able to change to Salbutamol/Albuterol MDI rescue for the duration of the study and judged capable of withholding albuterol/salbutamol for at least 6 hours prior to study visits.
* Subject must have their own Android or iPhone operating system (IOS) smart phone and a data package suitable for the installation and running of the app and sending and receiving data. Data used by the CIS is approximately 1 megabyte (MB) per month as a maximum; this is less data than a 1 minute video streamed from YouTube (2MB).
* Subjects must be willing and able to download the app on their personal smart phone and keep it turned on for the duration of the study. This will also require Bluetooth to be turned on for duration of the study. Subjects will also have to turn on mobile data for the app for the duration of study; unless travelling and when extra data roaming costs could be incurred.

Inclusion criteria for randomization:

* ACT score <20 at randomization visit (visit 2).

Exclusion Criteria:

* Subjects with a known or suspected alcohol or drug abuse which in the opinion of the investigator could interfere with the subject's proper completion of the protocol requirement.
* History of life threatening asthma: Defined as an asthma episode that required intubation and/or was associated with hypercapnea, respiratory arrest or hypoxic seizures within the last 6 months.
* A lower respiratory tract infection within 7 days of the screening visit.
* Concurrent diagnosis of chronic obstructive pulmonary disease (COPD) or other respiratory disorders including active tuberculosis, lung cancer, bronchiectasis, sarcoidosis, lung fibrosis, pulmonary hypertension, interstitial lung diseases or other active pulmonary diseases.
* History of hypersensitivity/intolerance to any components of the study inhalers (example, lactose, magnesium stearate). In addition, subjects with a history of severe milk protein allergy that, in the opinion of the study physician, contraindicates participation will also be excluded.
* Historical or current evidence of clinically significant or rapidly progressing or unstable cardiovascular, neurological, cardiovascular, neurological, renal, hepatic, immunological, endocrine (including uncontrolled diabetes or thyroid disease) or hematological abnormalities that are uncontrolled. Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the subject at risk through participation, or which would affect the analysis if the disease/condition exacerbated during the study.
* Subjects who have ever received treatment with biological based therapy example, omalizumab, mepolizumab, for asthma.
* Subjects who have received an investigational drug and/or medical device within 30 days of entry into this study (Screening), or within five drug half-lives of the investigational drug, whichever is longer.
* A subject will not be eligible for this study if he/she is an immediate family member of the participating investigator, sub-investigator, study coordinator, employee of the participating investigator, or any family member of a Propeller Health employee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 437 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2019-01-24 (Actual); Study Completion 2019-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (56):
- United States (11):
  - GSK Investigational Site, Aventura, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Flossmoor, Illinois
  - GSK Investigational Site, Glenview, Illinois
  - GSK Investigational Site, Hazelwood, Missouri
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Greenfield, Wisconsin
- Canada (12):
  - GSK Investigational Site, Kelowna, British Columbia
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Ajax, Ontario
  - GSK Investigational Site, Burlington, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Sarnia, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Windsor, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
  - GSK Investigational Site, Victoriaville, Quebec
- Germany (6):
  - GSK Investigational Site, Rüdersdorf, Brandenburg
  - GSK Investigational Site, Darmstadt, Hesse
  - GSK Investigational Site, Warendorf, North Rhine-Westphalia
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Berlin
- Italy (5):
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Salerno, Campania
  - GSK Investigational Site, Pordenone, Friuli Venezia Giulia
  - GSK Investigational Site, Palermo, Sicily
  - GSK Investigational Site, Pisa, Tuscany
- Netherlands (6):
  - GSK Investigational Site, Breda
  - GSK Investigational Site, Groningen
  - GSK Investigational Site, Hengelo
  - GSK Investigational Site, Hoorn
  - GSK Investigational Site, The Hague
  - GSK Investigational Site, Zutphen
- Spain (7):
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Balenyà (Barcelona)
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, La Roca Del Valles (Barcelona)
  - GSK Investigational Site, Loja/ Granada
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Peralada( Girona)
- United Kingdom (9):
  - GSK Investigational Site, Aylesbury, Buckinghamshire
  - GSK Investigational Site, Wigan, Lancashire
  - GSK Investigational Site, Wellingborough, Northamptonshire
  - GSK Investigational Site, Addlestone, Surrey
  - GSK Investigational Site, Rotherham, Yorkshire
  - GSK Investigational Site, Bristol
  - GSK Investigational Site, Chelmsford
  - GSK Investigational Site, Chertsey, Surrey
  - GSK Investigational Site, Harrogate

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20790

REFERENCES:
- [Derived] Moore A, Preece A, Sharma R, Heaney LG, Costello RW, Wise RA, Ludwig-Sengpiel A, Mosnaim G, Rees J, Tomlinson R, Tal-Singer R, Stempel DA, Barnes N. A randomised controlled trial of the effect of a connected inhaler system on medication adherence in uncontrolled asthmatic patients. Eur Respir J. 2021 Jun 4;57(6):2003103. doi: 10.1183/13993003.03103-2020. Print 2021 Jun. PMID 33334936

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label, randomized, multi-center, parallel group study to evaluate the effect of the connected inhaler system (CIS) on adherence to Relvar/Breo ELLIPTA therapy, in asthmatic participants (Par) with poor control.
Pre-assignment Details: A total of 528 participants were screened and 437 participants were enrolled and randomized in this study.
Groups:
- Cohort 1: Data on Maintenance Use Supplied to Par and HCP: Eligible participants received Relvar/Breo maintenance therapy at doses of 100/25 microgram (mcg) or 200/25 mcg per actuation administered via ELLIPTA dry powder inhaler (DPI), one inhalation once daily. Participants also received salbutamol rescue medication at dose of 100 mcg per actuation administered via metered dose inhaler (MDI), as and when required. Sensors were attached to both the inhalers to electronically record actuation data. Information from sensor attached to Relvar/Breo ELLIPTA was fed back to the participant via an application on smart phone and to the participant's healthcare professional (HCP) via an online dashboard.
- Cohort 2: Data on Maintenance Use Supplied to Par: Eligible participants received Relvar/Breo maintenance therapy at doses of 100/25 mcg or 200/25 mcg per actuation administered via ELLIPTA DPI, one inhalation once daily. Participants also received salbutamol rescue medication at dose of 100 mcg per actuation administered via MDI, as and when required. Sensors were attached to both the inhalers to electronically record actuation data. Information from sensor attached to Relvar/Breo ELLIPTA was fed back to the participant only via an application on smart phone.
- Cohort 3: Data on Maintenance and Rescue Use to Par and HCP: Eligible participants received Relvar/Breo maintenance therapy at doses of 100/25 mcg or 200/25 mcg per actuation administered via ELLIPTA DPI, one inhalation once daily. Participants also received salbutamol rescue medication at dose of 100 mcg per actuation administered via MDI, as and when required. Sensors were attached to both the inhalers to electronically record actuation data. Information from sensors attached to Relvar/Breo ELLIPTA and salbutamol MDI was fed back to the participant via an application on smart phone and to HCP via an online dashboard.
- Cohort 4: Data on Maintenance and Rescue Use Supplied to Par: Eligible participants received Relvar/Breo maintenance therapy at doses of 100/25 mcg or 200/25 mcg per actuation administered via ELLIPTA DPI, one inhalation once daily. Participants also received salbutamol rescue medication at dose of 100 mcg per actuation administered via MDI, as and when required. Sensors were attached to both the inhalers to electronically record actuation data. Information from sensors attached to Relvar/Breo ELLIPTA and salbutamol MDI was fed back to the participant via an application on smart phone.
- Cohort 5: No Data Supplied to Par or HCP: Eligible participants received Relvar/Breo maintenance therapy at doses of 100/25 mcg or 200/25 mcg per actuation administered via ELLIPTA DPI, one inhalation once daily. Participants also received salbutamol rescue medication at dose of 100 mcg per actuation administered via MDI, as and when required. Sensors were attached to both the inhalers to electronically record actuation data. Participants were provided with a home hub through which their data was uploaded during the study but the participants and their HCP were not able to view the data.
Period: Overall Study
Arm/Group | Cohort 1: Data on Maintenance Use Supplied to Par and HCP | Cohort 2: Data on Maintenance Use Supplied to Par | Cohort 3: Data on Maintenance and Rescue Use to Par and HCP | Cohort 4: Data on Maintenance and Rescue Use Supplied to Par | Cohort 5: No Data Supplied to Par or HCP
Started | 87 | 88 | 88 | 88 | 86
Completed | 82 | 81 | 77 | 78 | 81
Not Completed | 5 | 7 | 11 | 10 | 5
Not completed — Physician Decision | 0 | 1 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 3 | 3 | 5 | 2 | 1
Not completed — Lost to Follow-up | 0 | 2 | 4 | 3 | 1
Not completed — Protocol Violation | 1 | 0 | 1 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 2 | 1
Not completed — Adverse Event | 1 | 1 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Data on Maintenance Use Supplied to Par and HCP | Cohort 2: Data on Maintenance Use Supplied to Par | Cohort 3: Data on Maintenance and Rescue Use to Par and HCP | Cohort 4: Data on Maintenance and Rescue Use Supplied to Par | Cohort 5: No Data Supplied to Par or HCP | Total
Number analyzed (Participants) | 87 | 88 | 88 | 88 | 86 | 437
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.7 (15.79) | 47.0 (14.70) | 47.8 (15.28) | 47.8 (13.23) | 47.2 (15.91) | 47.3 (14.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 54 | 59 | 60 | 47 | 284
  Male | 23 | 34 | 29 | 28 | 39 | 153
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian (AI) or Alaska native (AN) | 1 | 0 | 0 | 0 | 2 | 3
  Asian-Central/South Asian Heritage | 1 | 3 | 1 | 2 | 1 | 8
  Asian-East Asian Heritage | 1 | 0 | 0 | 0 | 1 | 2
  Asian-South East (SE) Asian Heritage (AH) | 2 | 2 | 3 | 2 | 3 | 12
  Black or African American | 10 | 3 | 8 | 9 | 4 | 34
  Native Hawaiian or other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 1
  White-Arabic/North African heritage | 0 | 0 | 0 | 1 | 1 | 2
  White-White/Caucasian/European Heritage (EH) | 72 | 76 | 76 | 74 | 73 | 371
  AI or AN and Black or African American | 0 | 2 | 0 | 0 | 0 | 2
  AI or AN and White- White/Caucasian/EH | 0 | 1 | 0 | 0 | 0 | 1
  Asian-SE AH and White- White/Caucasian/EH | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of ELLIPTA Doses Taken (Daily Adherence) Between Month 4 and Month 6 as Determined by the Maintenance Sensor for Arms; ("Cohort 1: Data on Maintenance Use Supplied to Participant and HCP" and"Cohort 5: no Data Supplied to Participant or HCP")
Description: Daily adherence is defined as the participant taking one dose of Relvar/Breo ELLIPTA, within a 24-hour period, starting at 12.00 anti-meridiem (a.m.) each day of the treatment period. The percentage of ELLIPTA doses taken were determined by the clip-on sensor attached to ELLIPTA, which records the time and date when the ELLIPTA cover was opened and closed. Analysis was carried out by Analysis of Covariance (ANCOVA) model. Least Square mean percentage of ELLIPTA doses taken (daily adherence) between Months 4 and 6 was determined by the maintenance sensor daily adherence over the last three months of the study period (between months 4 to 6). The daily adherence to ELLIPTA maintenance therapy when both the participant and the HCP were supplied with data from the maintenance sensor (Cohort 1) versus no data supplied to the participant or HCP (Cohort 5) is summarized.
Time Frame: Month 4 to Month 6
Population: Intent-to-Treat (ITT) Population comprised of all randomized participants, excluding those who were randomized in error. Only those participants with adherence data observed/imputed at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of ELLIPTA doses
Arm/Group | Cohort 1: Data on Maintenance Use Supplied to Par and HCP | Cohort 5: No Data Supplied to Par or HCP
Number analyzed (Participants) | 83 | 85
Percentage of ELLIPTA doses | 80.9 (3.19) | 69.0 (3.19)
Statistical Analysis 1: Comparison: Cohort 1: Data on Maintenance Use Supplied to Par and HCP vs Cohort 5: No Data Supplied to Par or HCP; Test type: Superiority; p < 0.001, ANCOVA — p-value was calculated using ANCOVA; Mean Difference (Final Values) = 12.0, 95% CI 2-sided [5.2 to 18.8] — Analysis was performed by ANCOVA adjusted for randomized treatment arm, Baseline adherence, duration of run-in (visits), country, gender and age

2. Secondary Outcome: Percentage of ELLIPTA Doses Taken (Daily Adherence) Between Month 4 and Month 6 as Determined by the Maintenance Sensor
Description: Daily adherence is defined as the participant taking one dose of Relvar/Breo ELLIPTA, within a 24-hour period, starting at 12.00 a.m. each day of the treatment period. The percentage of ELLIPTA doses taken were determined by the clip-on sensor attached to ELLIPTA, which records the time and date when the ELLIPTA cover was opened and closed. Least Square mean percentage of ELLIPTA doses taken (daily adherence) between Months 4 and 6 was determined by the maintenance sensor daily adherence over the last three months of the study period (between months 4 to 6). The effect on daily adherence to maintenance therapy when maintenance data was only supplied to participants (Cohort 2), rescue and maintenance data were supplied to participant and HCP (Cohort 3), and rescue and maintenance data only supplied to participant (Cohort 4) versus no data supplied to the participant or HCP (Cohort 5) is summarized.
Time Frame: Month 4 to Month 6
Population: ITT Population. Only those participants with adherence data observed/imputed at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of ELLIPTA doses
Arm/Group | Cohort 2: Data on Maintenance Use Supplied to Par | Cohort 3: Data on Maintenance and Rescue Use to Par and HCP | Cohort 4: Data on Maintenance and Rescue Use Supplied to Par | Cohort 5: No Data Supplied to Par or HCP
Number analyzed (Participants) | 84 | 84 | 82 | 85
Percentage of ELLIPTA doses | 77.2 (3.04) | 78.3 (3.11) | 77.1 (3.25) | 69.0 (3.19)
Statistical Analysis 1: Comparison: Cohort 2: Data on Maintenance Use Supplied to Par vs Cohort 5: No Data Supplied to Par or HCP; Test type: Other; p = 0.016, ANCOVA — p-value was calculated using ANCOVA; Mean Difference (Final Values) = 8.2, 95% CI 2-sided [1.6 to 14.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohort 3: Data on Maintenance and Rescue Use to Par and HCP vs Cohort 5: No Data Supplied to Par or HCP; Test type: Other; p = 0.006, ANCOVA — p-value was calculated using ANCOVA; Mean Difference (Final Values) = 9.3, 95% CI 2-sided [2.7 to 16.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohort 4: Data on Maintenance and Rescue Use Supplied to Par vs Cohort 5: No Data Supplied to Par or HCP; Test type: Other; p = 0.018, ANCOVA — p-value was calculated using ANCOVA; Mean Difference (Final Values) = 8.1, 95% CI 2-sided [1.4 to 14.8] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Percentage of ELLIPTA Doses Taken (Daily Adherence) Between Month 1 and Month 3 as Determined by the Maintenance Sensor
Description: Daily adherence is defined as the participant taking one dose of Relvar/Breo ELLIPTA, within a 24-hour period, starting at 12.00 a.m. each day of the treatment period. The percentage of ELLIPTA doses taken were determined by the clip-on sensor attached to ELLIPTA, which records the time and date when the ELLIPTA cover was opened and closed. Least Square mean percentage of ELLIPTA doses taken (daily adherence) between Months 1 and 3 was determined by the maintenance sensor daily adherence. The effect on daily adherence to maintenance therapy when maintenance data was supplied to both the participant and the HCP (Cohort 1), maintenance data was only supplied to participants (Cohort 2), rescue and maintenance data were supplied to participant and HCP (Cohort 3), and rescue and maintenance data only supplied to participant (Cohort 4) versus no data supplied to the participant or HCP (Cohort 5) is summarized.
Time Frame: Month 1 to Month 3
Population: ITT Population. Only those participants with adherence data observed/imputed at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of ELLIPTA doses
Arm/Group | Cohort 1: Data on Maintenance Use Supplied to Par and HCP | Cohort 2: Data on Maintenance Use Supplied to Par | Cohort 3: Data on Maintenance and Rescue Use to Par and HCP | Cohort 4: Data on Maintenance and Rescue Use Supplied to Par | Cohort 5: No Data Supplied to Par or HCP
Number analyzed (Participants) | 86 | 87 | 88 | 88 | 86
Percentage of ELLIPTA doses | 85.7 (2.82) | 84.2 (2.66) | 82.0 (2.74) | 79.2 (2.78) | 76.4 (2.82)
Statistical Analysis 1: Comparison: Cohort 1: Data on Maintenance Use Supplied to Par and HCP vs Cohort 5: No Data Supplied to Par or HCP; Test type: Other; p = 0.003, ANCOVA — p-value was calculated using ANCOVA; Mean Difference (Final Values) = 9.3, 95% CI 2-sided [3.2 to 15.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohort 2: Data on Maintenance Use Supplied to Par vs Cohort 5: No Data Supplied to Par or HCP; Test type: Other; p = 0.011, ANCOVA — p-value was calculated using ANCOVA; Mean Difference (Final Values) = 7.7, 95% CI 2-sided [1.8 to 13.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohort 3: Data on Maintenance and Rescue Use to Par and HCP vs Cohort 5: No Data Supplied to Par or HCP; Test type: Other; p = 0.066, ANCOVA — p-value was calculated using ANCOVA; Mean Difference (Final Values) = 5.5, 95% CI 2-sided [-0.4 to 11.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Cohort 4: Data on Maintenance and Rescue Use Supplied to Par vs Cohort 5: No Data Supplied to Par or HCP; Test type: Other; p = 0.359, ANCOVA — p-value was calculated using ANCOVA; Mean Difference (Final Values) = 2.8, 95% CI 2-sided [-3.1 to 8.7] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Percentage of ELLIPTA Doses Taken (Daily Adherence) Between Month 1 and Month 6 as Determined by the Maintenance Sensor
Description: Daily adherence is defined as the participant taking one dose of Relvar/Breo ELLIPTA, within a 24-hour period, starting at 12.00 a.m. each day of the treatment period. The percentage of ELLIPTA doses taken were determined by the clip-on sensor attached to ELLIPTA, which records the time and date when the ELLIPTA cover was opened and closed. Least Square mean percentage of ELLIPTA doses taken (daily adherence) between Months 1 and 6 was determined by the maintenance sensor daily adherence. The effect on daily adherence to maintenance therapy when maintenance data was supplied to both the participant and the HCP (Cohort 1), maintenance data was only supplied to participants (Cohort 2), rescue and maintenance data were supplied to participant and HCP (Cohort 3), and rescue and maintenance data only supplied to participant (Cohort 4) versus no data supplied to the participant or HCP (Cohort 5) is summarized.
Time Frame: Month 1 to Month 6
Population: ITT Population. Only those participants with adherence data observed/imputed at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of ELLIPTA doses
Arm/Group | Cohort 1: Data on Maintenance Use Supplied to Par and HCP | Cohort 2: Data on Maintenance Use Supplied to Par | Cohort 3: Data on Maintenance and Rescue Use to Par and HCP | Cohort 4: Data on Maintenance and Rescue Use Supplied to Par | Cohort 5: No Data Supplied to Par or HCP
Number analyzed (Participants) | 86 | 87 | 88 | 88 | 86
Percentage of ELLIPTA doses | 81.5 (3.07) | 78.8 (2.90) | 77.7 (2.99) | 75.2 (3.03) | 71.8 (3.07)
Statistical Analysis 1: Comparison: Cohort 1: Data on Maintenance Use Supplied to Par and HCP vs Cohort 5: No Data Supplied to Par or HCP; Test type: Other; p = 0.004, ANCOVA — p-value was calculated using ANCOVA; Mean Difference (Final Values) = 9.7, 95% CI 2-sided [3.1 to 16.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohort 2: Data on Maintenance Use Supplied to Par vs Cohort 5: No Data Supplied to Par or HCP; Test type: Other; p = 0.032, ANCOVA — p-value was calculated using ANCOVA; Mean Difference (Final Values) = 7.1, 95% CI 2-sided [0.6 to 13.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohort 3: Data on Maintenance and Rescue Use to Par and HCP vs Cohort 5: No Data Supplied to Par or HCP; Test type: Other; p = 0.070, ANCOVA — p-value was calculated using ANCOVA; Mean Difference (Final Values) = 5.9, 95% CI 2-sided [-0.5 to 12.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Cohort 4: Data on Maintenance and Rescue Use Supplied to Par vs Cohort 5: No Data Supplied to Par or HCP; Test type: Other; p = 0.294, ANCOVA — p-value was calculated using ANCOVA; Mean Difference (Final Values) = 3.4, 95% CI 2-sided [-3.0 to 9.9] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Percentage of Rescue Free Days Between Month 4 and Month 6 as Determined by the Rescue Medication Sensor
Description: Data for rescue medication use was collected by the clip-on sensor for salbutamol MDI which records time and date when the MDI was actuated. Percentage of rescue free days were determined by the rescue sensor records of date, time and number of inhaler actuations. Least Square mean percentage of rescue free days between Months 4 and 6 when maintenance data was supplied to both the participant and the HCP (Cohort 1); maintenance data was only supplied to participants (Cohort 2); rescue and maintenance data were supplied to participant and HCP (Cohort 3) and rescue and maintenance data only supplied to participant (Cohort 4) versus no data supplied to the participant or HCP (Cohort 5) is summarized.
Time Frame: Month 4 to Month 6
Population: ITT Population. Only those participants with rescue data observed/imputed at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of rescue free days
Arm/Group | Cohort 1: Data on Maintenance Use Supplied to Par and HCP | Cohort 2: Data on Maintenance Use Supplied to Par | Cohort 3: Data on Maintenance and Rescue Use to Par and HCP | Cohort 4: Data on Maintenance and Rescue Use Supplied to Par | Cohort 5: No Data Supplied to Par or HCP
Number analyzed (Participants) | 87 | 88 | 88 | 88 | 85
Percentage of rescue free days | 81.1 (2.82) | 81.2 (2.66) | 85.6 (2.76) | 83.7 (2.80) | 76.4 (2.82)
Statistical Analysis 1: Comparison: Cohort 1: Data on Maintenance Use Supplied to Par and HCP vs Cohort 5: No Data Supplied to Par or HCP; Test type: Other; p = 0.118, ANCOVA — p-value was calculated using ANCOVA; Mean Difference (Final Values) = 4.8, 95% CI 2-sided [-1.2 to 10.8] — Analysis was performed by ANCOVA adjusted for randomized treatment arm, Baseline rescue use, duration of run-in (visits), country, gender and age
Statistical Analysis 2: Comparison: Cohort 2: Data on Maintenance Use Supplied to Par vs Cohort 5: No Data Supplied to Par or HCP; Test type: Other; p = 0.105, ANCOVA — p-value was calculated using ANCOVA; Mean Difference (Final Values) = 4.8, 95% CI 2-sided [-1.0 to 10.7] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Cohort 3: Data on Maintenance and Rescue Use to Par and HCP vs Cohort 5: No Data Supplied to Par or HCP; Test type: Other; p = 0.002, ANCOVA — p-value was calculated using ANCOVA; Mean Difference (Final Values) = 9.2, 95% CI 2-sided [3.3 to 15.1] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: Cohort 4: Data on Maintenance and Rescue Use Supplied to Par vs Cohort 5: No Data Supplied to Par or HCP; Test type: Other; p = 0.015, ANCOVA — p-value was calculated using ANCOVA; Mean Difference (Final Values) = 7.3, 95% CI 2-sided [1.5 to 13.2] — [estimate comment as in outcome 5, analysis 1]

6. Secondary Outcome: Number of Doses of Rescue Medication Use Between Month 4 and Month 6 as Determined by the Rescue Medication Sensor
Description: Data for rescue medication use was collected by the clip-on sensor for salbutamol MDI which records time and date when the MDI was actuated. Total rescue use was determined by the rescue sensor records of date, time and number of inhaler actuations. The mean number of doses of rescue medicines between Months 4 and 6 when maintenance data was supplied to both the participant and the HCP (Cohort 1); maintenance data was only supplied to participants (Cohort 2); rescue and maintenance data were supplied to participant and HCP (Cohort 3) and rescue and maintenance data only supplied to participant (Cohort 4) versus no data supplied to the participant or HCP (Cohort 5) is summarized.
Time Frame: Month 4 to Month 6
Population: ITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Doses of rescue medication
Arm/Group | Cohort 1: Data on Maintenance Use Supplied to Par and HCP | Cohort 2: Data on Maintenance Use Supplied to Par | Cohort 3: Data on Maintenance and Rescue Use to Par and HCP | Cohort 4: Data on Maintenance and Rescue Use Supplied to Par | Cohort 5: No Data Supplied to Par or HCP
Number analyzed (Participants) | 83 | 84 | 85 | 82 | 85
Doses of rescue medication | 55.3 (107.73) | 40.6 (91.53) | 29.5 (54.41) | 27.0 (45.27) | 55.8 (158.49)

7. Secondary Outcome: Change From Baseline in Asthma Control Test (ACT) Total Score
Description: The ACT is a validated self-completed questionnaire utilizing 5 questions to assess asthma control on a 5-point categorical scale ranging from 1 (not controlled at all) to 5 (completely controlled). Total score is calculated as the sum of the scores from the 5 questions and can range from 5 to 25, with higher scores indicating better control. An ACT total score of 5 to 19 suggests that the participant's asthma is unlikely to be well controlled, whilst a score of 20 to 25 suggests that the participant's asthma is likely to be well controlled. Baseline value was the latest assessment prior to randomization (Day 1, pre-dose). Change from Baseline was calculated as post-dose visit value minus the Baseline value.
Time Frame: Baseline and Month 6
Population: ITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Cohort 1: Data on Maintenance Use Supplied to Par and HCP | Cohort 2: Data on Maintenance Use Supplied to Par | Cohort 3: Data on Maintenance and Rescue Use to Par and HCP | Cohort 4: Data on Maintenance and Rescue Use Supplied to Par | Cohort 5: No Data Supplied to Par or HCP
Number analyzed (Participants) | 82 | 82 | 78 | 78 | 82
Scores on a Scale | 3.4 (0.40) | 4.3 (0.40) | 4.7 (0.41) | 4.2 (0.41) | 3.9 (0.40)
Statistical Analysis 1: Comparison: Cohort 1: Data on Maintenance Use Supplied to Par and HCP vs Cohort 5: No Data Supplied to Par or HCP; Test type: Other; p = 0.400, MMRM — p-value was calculated using Mixed Model Repeated Measures (MMRM); Mean Difference (Net) = -0.5, 95% CI 2-sided [-1.6 to 0.6] — Analysis was performed by MMRM adjusted for randomized treatment arm,Baseline ACT total score,randomized treatment arm-by-visit interaction,Baseline ACT total score-by-visit interaction,gender,age,country and participant fitted as a random factor
Statistical Analysis 2: Comparison: Cohort 2: Data on Maintenance Use Supplied to Par vs Cohort 5: No Data Supplied to Par or HCP; Test type: Other; p = 0.441, MMRM — p-value was calculated using MMRM; Mean Difference (Net) = 0.4, 95% CI 2-sided [-0.7 to 1.5] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 3: Comparison: Cohort 3: Data on Maintenance and Rescue Use to Par and HCP vs Cohort 5: No Data Supplied to Par or HCP; Test type: Other; p = 0.164, MMRM — p-value was calculated using MMRM; Mean Difference (Net) = 0.8, 95% CI 2-sided [-0.3 to 1.9] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 4: Comparison: Cohort 4: Data on Maintenance and Rescue Use Supplied to Par vs Cohort 5: No Data Supplied to Par or HCP; Test type: Other; p = 0.661, MMRM — p-value was calculated using MMRM; Mean Difference (Net) = 0.3, 95% CI 2-sided [-0.9 to 1.4] — [estimate comment as in outcome 7, analysis 1]

8. Secondary Outcome: Percentage of Participants Attaining Asthma Control (Percentage of Participants With an ACT Total Score >=20) at Month 6
Description: Percentage of participants attaining asthma control was defined as participants with an ACT total score >=20 at Month 6. The ACT is a validated self-completed questionnaire utilizing 5 questions to assess asthma control on a 5-point categorical scale ranging from 1 (not controlled at all) to 5 (completely controlled). Total score is calculated as the sum of the scores from the 5 questions and can range from 5 to 25, with higher scores indicating better control. An ACT total score of 5 to 19 suggests that the participant's asthma is unlikely to be well controlled, whilst a score of 20 to 25 suggests that the participant's asthma is likely to be well controlled. Percentage of participants who attained asthma control at Month 6 is presented.
Time Frame: Month 6
Population: ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1: Data on Maintenance Use Supplied to Par and HCP | Cohort 2: Data on Maintenance Use Supplied to Par | Cohort 3: Data on Maintenance and Rescue Use to Par and HCP | Cohort 4: Data on Maintenance and Rescue Use Supplied to Par | Cohort 5: No Data Supplied to Par or HCP
Number analyzed (Participants) | 87 | 88 | 88 | 88 | 86
Percentage of participants | 52 | 66 | 55 | 53 | 62
Statistical Analysis 1: Comparison: Cohort 1: Data on Maintenance Use Supplied to Par and HCP vs Cohort 5: No Data Supplied to Par or HCP; Test type: Other; p = 0.385, Regression, Logistic — p-value was calculated using logistic regression; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.39 to 1.44] — Analysis was performed by logistic regression adjusted for randomized treatment arm, Baseline ACT total score, country, gender and age
Statistical Analysis 2: Comparison: Cohort 2: Data on Maintenance Use Supplied to Par vs Cohort 5: No Data Supplied to Par or HCP; Test type: Other; p = 0.517, Regression, Logistic — p-value was calculated using logistic regression; Odds Ratio (OR) = 1.24, 95% CI 2-sided [0.64 to 2.42] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Cohort 3: Data on Maintenance and Rescue Use to Par and HCP vs Cohort 5: No Data Supplied to Par or HCP; Test type: Other; p = 0.921, Regression, Logistic — p-value was calculated using logistic regression; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.51 to 1.85] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 4: Comparison: Cohort 4: Data on Maintenance and Rescue Use Supplied to Par vs Cohort 5: No Data Supplied to Par or HCP; Test type: Other; p = 0.321, Regression, Logistic — p-value was calculated using logistic regression; Odds Ratio (OR) = 0.72, 95% CI 2-sided [0.38 to 1.38] — [estimate comment as in outcome 8, analysis 1]

9. Secondary Outcome: Percentage of Participants With an Increase From Baseline >=3 in ACT Total Score at Month 6
Description: The ACT is a validated self-completed questionnaire utilizing 5 questions to assess asthma control on a 5-point categorical scale ranging from 1 (not controlled at all) to 5 (completely controlled). Total score is calculated as the sum of the scores from the 5 questions and can range from 5 to 25, with higher scores indicating better control. An ACT total score of 5 to 19 suggests that the participant's asthma is unlikely to be well controlled, whilst a score of 20 to 25 suggests that the participant's asthma is likely to be well controlled. Baseline value was the latest assessment prior to randomization (Day 1, pre-dose). Percentage of participants with an increase from Baseline >=3 in ACT total score at Month 6 is presented.
Time Frame: Baseline and Month 6
Population: ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1: Data on Maintenance Use Supplied to Par and HCP | Cohort 2: Data on Maintenance Use Supplied to Par | Cohort 3: Data on Maintenance and Rescue Use to Par and HCP | Cohort 4: Data on Maintenance and Rescue Use Supplied to Par | Cohort 5: No Data Supplied to Par or HCP
Number analyzed (Participants) | 87 | 88 | 88 | 88 | 86
Percentage of participants | 61 | 69 | 65 | 63 | 64
Statistical Analysis 1: Comparison: Cohort 1: Data on Maintenance Use Supplied to Par and HCP vs Cohort 5: No Data Supplied to Par or HCP; Test type: Other; p = 0.911, Regression, Logistic — p-value was calculated using logistic regression; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.54 to 1.98] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: Cohort 2: Data on Maintenance Use Supplied to Par vs Cohort 5: No Data Supplied to Par or HCP; Test type: Other; p = 0.383, Regression, Logistic — p-value was calculated using logistic regression; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.70 to 2.54] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Cohort 3: Data on Maintenance and Rescue Use to Par and HCP vs Cohort 5: No Data Supplied to Par or HCP; Test type: Other; p = 0.814, Regression, Logistic — p-value was calculated using logistic regression; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.57 to 2.04] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 4: Comparison: Cohort 4: Data on Maintenance and Rescue Use Supplied to Par vs Cohort 5: No Data Supplied to Par or HCP; Test type: Other; p = 0.986, Regression, Logistic — p-value was calculated using logistic regression; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.53 to 1.89] — [estimate comment as in outcome 8, analysis 1]

10. Secondary Outcome: Percentage of Participants Who Have Either an ACT Total Score of >=20 and/or an Increase From Baseline >=3 in ACT Total Score at Month 6
Description: The ACT is a validated self-completed questionnaire utilizing 5 questions to assess asthma control on a 5-point categorical scale ranging from 1 (not controlled at all) to 5 (completely controlled). Total score is calculated as the sum of the scores from the 5 questions and can range from 5 to 25, with higher scores indicating better control. Baseline value was the latest assessment prior to randomization (Day 1, pre-dose). Percentage of participants who had either an ACT total score of >=20 and/or an increase from Baseline >=3 in ACT total score at Month 6 is presented.
Time Frame: Baseline and Month 6
Population: ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1: Data on Maintenance Use Supplied to Par and HCP | Cohort 2: Data on Maintenance Use Supplied to Par | Cohort 3: Data on Maintenance and Rescue Use to Par and HCP | Cohort 4: Data on Maintenance and Rescue Use Supplied to Par | Cohort 5: No Data Supplied to Par or HCP
Number analyzed (Participants) | 87 | 88 | 88 | 88 | 86
Percentage of participants | 66 | 75 | 65 | 67 | 70
Statistical Analysis 1: Comparison: Cohort 1: Data on Maintenance Use Supplied to Par and HCP vs Cohort 5: No Data Supplied to Par or HCP; Test type: Other; p = 0.833, Regression, Logistic — p-value was calculated using logistic regression; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.48 to 1.81] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: Cohort 2: Data on Maintenance Use Supplied to Par vs Cohort 5: No Data Supplied to Par or HCP; Test type: Other; p = 0.383, Regression, Logistic — p-value was calculated using logistic regression; Odds Ratio (OR) = 1.35, 95% CI 2-sided [0.69 to 2.67] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Cohort 3: Data on Maintenance and Rescue Use to Par and HCP vs Cohort 5: No Data Supplied to Par or HCP; Test type: Other; p = 0.628, Regression, Logistic — p-value was calculated using logistic regression; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.44 to 1.63] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 4: Comparison: Cohort 4: Data on Maintenance and Rescue Use Supplied to Par vs Cohort 5: No Data Supplied to Par or HCP; Test type: Other; p = 0.844, Regression, Logistic — p-value was calculated using logistic regression; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.49 to 1.80] — [estimate comment as in outcome 8, analysis 1]

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the start of study treatment up to 6 months
Description: SAEs and non-serious AEs were reported for the ITT Population which comprised of all randomized participants, excluding those who were randomized in error.
Arm/Group | Cohort 1: Data on Maintenance Use Supplied to Par and HCP | Cohort 2: Data on Maintenance Use Supplied to Par | Cohort 3: Data on Maintenance and Rescue Use to Par and HCP | Cohort 4: Data on Maintenance and Rescue Use Supplied to Par | Cohort 5: No Data Supplied to Par or HCP
All-Cause Mortality (participants affected / at risk) | 0/87 | 0/88 | 0/88 | 0/88 | 0/86
Serious Adverse Events (participants affected / at risk) | 2/87 | 1/88 | 2/88 | 1/88 | 4/86
Other Adverse Events (participants affected / at risk) | 4/87 | 1/88 | 1/88 | 1/88 | 2/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Data on Maintenance Use Supplied to Par and HCP (N=87) | Cohort 2: Data on Maintenance Use Supplied to Par (N=88) | Cohort 3: Data on Maintenance and Rescue Use to Par and HCP (N=88) | Cohort 4: Data on Maintenance and Rescue Use Supplied to Par (N=88) | Cohort 5: No Data Supplied to Par or HCP (N=86)
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Obstructive pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Ovarian germ cell teratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Data on Maintenance Use Supplied to Par and HCP (N=87) | Cohort 2: Data on Maintenance Use Supplied to Par (N=88) | Cohort 3: Data on Maintenance and Rescue Use to Par and HCP (N=88) | Cohort 4: Data on Maintenance and Rescue Use Supplied to Par (N=88) | Cohort 5: No Data Supplied to Par or HCP (N=86)
Oral candidiasis (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Oral fungal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-09-10): https://cdn.clinicaltrials.gov/large-docs/29/NCT03380429/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-21): https://cdn.clinicaltrials.gov/large-docs/29/NCT03380429/SAP_001.pdf